CLINICAL TRIAL: NCT02994654
Title: CONTINUED ACCESS PROTOCOL: Demonstration of the Safety and Effectiveness of ReCell® Combined With Meshed Skin Graft for Reduction of Donor Area in the Treatment of Acute Burn Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTP001-7
Record Dates: First submitted 2016-12-12; First posted 2016-12-16 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReCell (Experimental): All subjects will receive both ReCell and skin graft. Each patient serves as their own control. Their study treatment area (burn injury) will be divided into Area A and Area B. Investigational treatment will be randomly allocated to either Area A or Area B
  Interventions: Device: ReCell
- Control (Experimental): All subjects will receive both ReCell and skin graft. Each patient serves as their own control. Their study treatment area (burn injury) will be divided into Area A and Area B. Control, which is the Investigator's pre-determined graft plan will be randomly allocated to either Area A or Area B
  Interventions: Device: ReCell

INTERVENTIONS:
Device: ReCell — The ReCell-assigned treatment area will be treated as described in the product's Instructions for Use. In summary, 1ml of fluid physically covers a treatment area of 80 cm2. Each milliliter of fluid contains cells harvested from a square centimeter of thin split-thickness skin sample.
  The reagents and components of the ReCell kit are used, in a scalable fashion, to facilitate disaggregation of cells from skin samples into filtered cell suspension. Areas to be harvested for skin samples are to be clean and show no evidence of surrounding cellulitis or infection. Treatment area sizes and cell suspension volumes are to be recorded.

SUMMARY:
The overall purpose of this is study to provide continued access to the ReCell device following completion of protocol CTP001-6, and allow for collection of supplementary clinical outcome data for the ReCell device when used as an adjunct to meshed grafts in subjects with acute thermal burn injuries who require skin grafting for closure of burn injuries.

ELIGIBILITY:
Inclusion Criteria:

1. The subject requires skin grafting as a result of an acute thermal burn injury (i.e. injuries caused by exposure of the skin to fire/flames, excessive heat, hot steam or water).
2. The area of total burn injury is 5-50% TBSA inclusive.
3. Two areas requiring skin grafting, each at least 300cm2 (or 600cm2 contiguous), excluding hand/face and joints.
4. The subject is at least 5 years of age.
5. The subject (or family, for those under 18 years of age) is willing and able to complete all follow-up evaluations required by the study protocol.
6. The subject is to abstain from any other treatment of the wound(s) for the duration of the study unless medically necessary.
7. The subject agrees to abstain from enrollment in any other interventional clinical trial for the duration of the study.
8. The subject and/or guardian are able to read and understand instructions and give informed, voluntary, written consent.

Exclusion Criteria:

1. The subject's burn injuries were caused by chemicals, electricity, and/or radioactive substances.
2. The subject is unable to follow the protocol.
3. The subject has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives.
4. The subject has a known hypersensitivity to trypsin or compound sodium lactate for irrigation (Hartmann's) solution.
5. Life expectancy is less than 1year.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10; Primary Completion 2017-12 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Arizona Burn Center at Maricopa Integrated Health Systems, Phoenix, Arizona
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - U.S.Army Institute of Surgical Research, Fort Sam Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: All Participants (Within Patient Control): Every subject received both interventions (RECELL and CONTROL) such that each subject served as their own control. Each subject's study treatment area (burn injury) was divided into Area A and Area B before the areas (A and B) were randomly assigned to receive CONTROL (grafting consistent with the pre-identified graft plan) or RECELL (RECELL-generated cell suspension applied over a graft more widely meshed than identified in the pre-specified graft plan).
Period: Overall Study
Arm/Group | Experimental: All Participants (Within Patient Control)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: All Participants (Within Patient Control): All subjects receive both ReCell treatment and autograft (Area A and Area B). Each subject serves as their own control. Wound regions were randomly assigned to receive an autograft consistent with the investigator's pre-identified graft plan (Control) or to receive application of the ReCell-generated cell suspension over an autograft more widely meshed than identified in the investigator's pre-specified graft plan (ReCell-treated).
Arm/Group | Experimental: All Participants (Within Patient Control)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Confirmed Treatment Area Closure of RECELL-treated Wounds Compared to Control (Non-inferiority)
Description: Complete wound closure is defined as skin re-epithelialization without drainage, confirmed at two consecutive study visits at least 2 weeks apart by direct visualization by a qualified clinician blinded to treatment assignment. The incidence of complete wound closure is hypothesized to be non-inferior for ReCell-treated areas as compared to control areas.
Time Frame: Prior to or at 8 weeks
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Groups:
- ReCell: All subjects will receive both ReCell and skin graft. Each patient serves as their own control. Their study treatment area (burn injury) will be divided into Area A and Area B. Investigational treatment will be randomly allocated to either Area A or Area B
  ReCell: The ReCell-assigned treatment area will be treated as described in the product's Instructions for Use. In summary, 1ml of fluid physically covers a treatment area of 80 cm2. Each milliliter of fluid contains cells harvested from a square centimeter of thin split-thickness skin sample.
  The reagents and components of the ReCell kit are used, in a scalable fashion, to facilitate disaggregation of cells from skin samples into filtered cell suspension. Areas to be harvested for skin samples are to be clean and show no evidence of surrounding cellulitis or infection. Treatment area sizes and cell suspension volumes are to be recorded.
- Control: All subjects will receive both ReCell and skin graft. Each patient serves as their own control. Their study treatment area (burn injury) will be divided into Area A and Area B. Control, which is the Investigator's pre-determined graft plan will be randomly allocated to either Area A or Area B
  ReCell: The ReCell-assigned treatment area will be treated as described in the product's Instructions for Use. In summary, 1ml of fluid physically covers a treatment area of 80 cm2. Each milliliter of fluid contains cells harvested from a square centimeter of thin split-thickness skin sample.
  The reagents and components of the ReCell kit are used, in a scalable fashion, to facilitate disaggregation of cells from skin samples into filtered cell suspension. Areas to be harvested for skin samples are to be clean and show no evidence of surrounding cellulitis or infection. Treatment area sizes and cell suspension volumes are to be recorded.
Arm/Group | ReCell | Control
Number analyzed (Participants) | 9 | 9
Participants | 9 | 9

2. Primary Outcome: Relative Reduction in Donor Skin Area Requirement
Description: For this second co-primary endpoint, it is hypothesized that the expansion ratio associated with the RECELL treatment area will be superior to that of the control, i.e. less donor skin will be required for RECELL-treated areas compared with the control areas.
Time Frame: Prior to or at 8 weeks
Population: Intent-to-Treat Population
Measure: Geometric Mean (Standard Deviation); unit: cm2
Arm/Group | ReCell | Control
Number analyzed (Participants) | 12 | 12
cm2 | 2.1139 (2.2893) | 1.6523 (1.7578)

ADVERSE EVENTS:
Time Frame: 52 Weeks
Groups:
- All Participants: All subjects receive both ReCell treatment and autograft (Area A and Area B). Each subject serves as their own control. Wound regions were randomly assigned to receive an autograft consistent with the investigator's pre-identified graft plan (Control) or to receive application of the ReCell-generated cell suspension over an autograft more widely meshed than identified in the investigator's pre-specified graft plan (ReCell-treated).
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=12)
Failed Skin Graft (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Delayed Wound Healing (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Failed Skin Graft (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Respiratory Distress (Injury, poisoning and procedural complications) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=12)
Failed Skin Graft (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Delayed Wound Healing (General disorders) | 1 (1) — RECELL
Graft Loss Left Abdomen (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Non-healing Burn Wound (General disorders) | 1 (1) — RECELL
Severe Intermittent Nerve Pain (Vascular disorders) | 1 (1) — CONTROL
Graft Loss Right Abdomen (Injury, poisoning and procedural complications) | 1 (1) — CONTROL
Failed Skin Graft (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Right Thigh Graft Loss (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Graft Loss Left Upper Arm (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Hypertrophic Scar (Injury, poisoning and procedural complications) | 1 (1) — NON-STUDY AREA
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02994654/Prot_SAP_002.pdf